CLINICAL TRIAL: NCT04602715
Title: The Safety, Efficacy, and Tolerability of Microbial Ecosystem Therapeutic-2 in People With Major Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET-2 301-2
Record Dates: First submitted 2020-10-09; First posted 2020-10-26 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: two arm, randomized, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Hospital pharmacies will be provided with the randomization code and will dispense the appropriate medication to subjects. A fire-wall exists between the pharmacies and the investigational staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET-2 20 g (Experimental): Loading dose of MET-2 is administered for the first two days, followed by a regular, daily dose for the duration of the study (6 weeks total).The loading dose will consist of 5 g of MET-2 in the form of ten capsules orally on day one and on day two. The regular daily dose will consist of 1.5 g MET-2 in the form of three MET-2 capsules taken once daily, excluding days where they take the booster (same as loading dose).
  Interventions: Drug: MET-2
- Placebo (Placebo Comparator): Loading dose of placebo is administered for the first two days, followed by a regular, daily dose of placebo for the duration of the study (6 weeks total).The loading dose will consist of ten capsules of placebo (which match the MET-2 capsules in appearance and weight) taken orally on day one and on day two. The regular daily dose will consist of three placebo capsules taken once daily, excluding days where they take the booster (same as loading dose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MET-2 — Subjects will take capsules containing MET-2 daily during the trial. There will be a loading dose at the start of dosing, and a daily dose. There will be a booster dose given at week 2 and a second booster dose taken at week 4 for those subjects who have not improved by that time.
  Arms: MET-2 20 g
Drug: Placebo — Placebo Control
  Arms: Placebo

SUMMARY:
To measure the effects of Microbial Ecosystem Therapeutics (MET)-2 on symptoms of depression and anxiety using pre- and post-treatment scores for overall depression and anxiety

DETAILED DESCRIPTION:
An eight week, randomized, placebo controlled trial to assess subjective changes in mood and anxiety symptoms from baseline to after MET-2 treatment in participants with depression, using MADRS, Hamilton Anxiety Rating Scale (HAM-A), and other mood/anxiety scales and to demonstrate a significantly higher proportion of responders in patient who were randomized to receive the active study drug compared to patients who were randomized to receive placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent.
2. Not pregnant
3. Willing to participate in follow up as part of the study
4. Diagnosis of Major Depressive Disorder (MDD) by the Mini-International Neuropsychiatric Interview (MINI)
5. Current depressive episode with a Montgomery-Asberg Depression Rating Scale (MADRS) score of ≥15.
6. Able to understand and comply with the requirements of the study
7. Able to provide stool, urine, and blood samples.
8. Those who do not choose to use antidepressants for moderate-severe depression.

Exclusion Criteria:

1. History of chronic diarrhea
2. Need for regular use of agents that affect gastro-intestinal (GI) motility (narcotics such as codeine or morphine, agents such as loperamide or metoclopramide)
3. Colostomy
4. Elective surgery that will require preoperative antibiotics planned within 6 months of enrolment
5. History of bariatric surgery.
6. Pregnant, breastfeeding, or planning to get pregnant in the next 6 months
7. Any condition for which, in the opinion of the investigator, the participant should be excluded from the study.
8. Current use of any antidepressant/antianxiety drug (eligible to participate after a 4-week washout period)
9. More than three depressive episodes throughout lifetime
10. Having failed an anti-depressant treatment during current depressive episode
11. Use of any antibiotic drug in the past 4 weeks (may be eligible to participate after a 1-month washout period)
12. History of alcohol or substance dependence in the past 6 months
13. Daily use of probiotic product in the past 2 weeks (may be eligible to participate after a 2-week washout period)
14. Use of any type of laxative in the last 2 weeks.
15. Consumption of products fortified in probiotics (may be eligible to participate after a 2-week washout period)
16. High suicidal risk, as measured by MADRS item 10 score more than 3
17. Current psychotic symptoms
18. Bipolar Depression
19. History of epilepsy or uncontrolled seizures
20. Immunodeficiency (immuno-compromised and immuno-suppressed participants; e.g. acquired immune deficiency syndrome [AIDS], lymphoma, participants undergoing long-term corticosteroid treatment, chemotherapy and allograft participants)
21. Unstable medical conditions or serious diseases/conditions (e.g. cancer, cardiovascular, renal, lung, diabetes, psychiatric illness, bleeding disorders, etc.)
22. The use of natural health products (NHP); e.g. St. John's Wort, passion flower, etc.) that affect depression
23. History of Electroconvulsive therapy (ECT)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in Major Depression Symptoms | Baseline vs. Week 6
  To assess subjective changes in mood from baseline to after MET-2 treatment using the Montgomery-Asberg Depression Rating Scale (10 domains given a rating from 0 to 6)
Change in Anxiety Symptoms | Baseline vs. Week 6
  To assess subjective changes in anxiety symptoms from baseline to after MET-2 treatment using the Hamilton Anxiety Rating Scale (14 domains given a rating on a 5 point scale)

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, MD/PhD, Principal Investigator — Queens University
Locations (2):
- Canada (2):
  - Providence Care Hospital, Kingston, Ontario
  - CAMH, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chinna Meyyappan A, Sgarbossa C, Bromley H, Forth E, Muller DJ, Vazquez G, Cabrera C, Milev R. The Safety and Efficacy of Microbial Ecosystem Therapeutic-2 in People With Major Depression - A Phase 2, Double-Blind, Placebo-Controlled Study: Clinical Results: Innocuite et efficacite du traitement de l'ecosysteme microbien (met-2) dans la depression majeure - une etude de phase 2 a double insu controlee par placebo : resultats cliniques. Can J Psychiatry. 2025 Nov;70(11):816-823. doi: 10.1177/07067437251328270. Epub 2025 Mar 21. PMID 40116713
- [Derived] Chinna Meyyappan A, Sgarbossa C, Vazquez G, Bond DJ, Muller DJ, Milev R. The Safety and Efficacy of Microbial Ecosystem Therapeutic-2 in People With Major Depression: Protocol for a Phase 2, Double-Blind, Placebo-Controlled Study. JMIR Res Protoc. 2021 Sep 22;10(9):e31439. doi: 10.2196/31439. PMID 34550085